CLINICAL TRIAL: NCT00276640
Title: Cooperative Multicenter Study for Children and Adolescents With Low Grade Glioma
Brief Title: Radiation Therapy or Combination Chemotherapy in Treating Patients With Clinically or Radiologically Progressive Low-Grade Gliomas
Acronym: SIOP-LGG-2004
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Responsible Party: Principal Investigator, Astrid K. Gnekow, Chairlady, Societe Internationale d'Oncologie Pediatrique
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454506; 2005-005377-29 (EudraCT Number)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Primary Central Nervous System Neoplasms
Keywords: recurrent childhood brain stem glioma; untreated childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; untreated childhood cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; childhood oligodendroglioma; recurrent childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway and hypothalamic glioma; childhood spinal cord neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Optic Nerve Glioma; Spinal Cord Neoplasms | interventions — Vincristine; Carboplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vincristine, carboplatin (Active Comparator): standard chemotherapy group
  Interventions: Drug: vincristine, carboplatin
- vincristine, carboplatin, etoposide (Active Comparator): intensified induction chemotherapy group
  Interventions: Drug: vincristine, carboplatin, etoposide
- radiation (Active Comparator): radiation therapy group
  Interventions: Radiation: radiation therapy
- Control (No Intervention): Control group: wait and see strategy

INTERVENTIONS:
Drug: vincristine, carboplatin — vincristine: 1,5 mg/m² i.v., week 1,2,3,4,5,6,7,8,9,10,13,17,21
  carboplatin: 550 mg/m² i.v., week 1,4,7,10,13,17,21
  Arms: vincristine, carboplatin
Drug: vincristine, carboplatin, etoposide — vincristine: 1,5 mg/m² i.v., week 1,2,3,4,5,6,7,8,9,10,13,17,21
  carboplatin: 550 mg/m² i.v., week 1,4,7,10,13,17,21
  etoposide: 100 mg/m² i.v., week 1,4,7,10
  Arms: vincristine, carboplatin, etoposide
Radiation: radiation therapy — intracranial tumor site: 30 fractions, dose per fraction: 1.8 Gy, total dose: 54 Gy, duration 6 weeks
  spinal tumor site: 28 fractions, dose per fraction: 1.8 Gy, total dose: 50.4 Gy duration 5 1/2 weeks
  Arms: radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This clinical trial is studying giving radiation therapy or combination chemotherapy to see how well it works in treating patients with clinically or radiologically progressive low-grade gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide a comprehensive treatment strategy for children and adolescents with low-grade glioma of all tumour locations and histologies.
* Provide standardized treatment indication and treatment recommendations for non-surgical therapy in children and adolescents with low grade glioma without and with associated neurofibrosis-type 1 (NF1) at diagnosis or after observation.
* Determine overall, event-free, and progression-free survival.
* Radiotherapy arm: a. Determine progression free survival in older children without NF1 treated with radiotherapy using modern techniques for planning and treatment. b. Determine the reduction of the rate and intensity of possible late effects of therapy to the organs at risk by optimized planning and treatment.
* Chemotherapy arm: a. Determine progression free survival for younger children without NF1 treated with chemotherapy and randomized to either the 2-drug or the 3-drug induction regimen. b. Determine the distribution of response at week 24 (after induction) for younger children without NF1 treated with chemotherapy and randomized to either the 2-drug or the 3-drug induction regimen. c. Determine progression free survival for children with NF1treated with chemotherapy.
* Determine the influence of clinical and histological findings on overall survival, progression-free and event-free survival in these patients.
* Determine prospectively the late effects of tumor and therapy in these patients.

OUTLINE: This is a partially randomized, open-label, multicenter study.

Children with completely resected tumors, incompletely resected tumors, or those with clinically/neuroradiologically diagnosed tumors, who do not have severe symptoms at diagnosis, are only observed during follow-up.

Children with unresectable/incompletely-resectable tumors, or those with relapsed disease and those observed following incomplete initial resection or neuroradiologic diagnosis and clinical and/or neuro-radiologic progression receive non-surgical therapy. This non-surgical therapy is either chemotherapy (for children younger than 8 years and those with neurofibrosis-type 1 [NF1]) or radiotherapy (for children older than 8 years).

* Chemotherapy: Within the chemotherapy arm, patients without NF1 are randomized to receive 1 of 2 induction chemotherapy regimens. Patients with NF1 receive the two-drug induction therapy as in arm I.

  * Arm I (two-drug induction therapy [vincristine-carboplatin] ): Patients receive induction therapy comprising vincristine IV on day 1 of weeks 1-10 and weeks 13, 17, and 21 and carboplatin IV over 1 hour on day 1 of weeks 1, 4, 7, 10, 13, 17, and 21.
  * Arm II (three-drug induction therapy [vincristine-carboplatin-etoposide]): Patients receive vincristine and carboplatin as in two-drug induction therapy. Patients also receive etoposide IV over 1 hour on days 1-3 of weeks 1, 4, 7, and 10.

Beginning in week 25, all patients in the chemotherapy arm receive consolidation therapy comprising vincristine IV on days 1, 8, and 15 and carboplatin IV over 1 hour on day 1. Treatment repeats every 6 weeks for 9 courses. Patients experiencing disease progression or an allergic reaction to carboplatin receive vincristine IV on days 1, 8, and 15 and either cyclophosphamide IV over 1 hour on day 1 or cisplatin IV over 3 hours on days 1 and 2. Treatment repeats every 6 weeks for 5 courses. All patients in the chemotherapy arm receive a total of 18 months of treatment.

* Radiotherapy: Conventional external beam fractionated radiotherapy is given at standard doses for children receiving radiotherapy. Brachytherapy can be given, if tumors are suitable for this type of treatment.

After completion of study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 520 patients will be accrued for the randomized arm of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade glioma, of 1 of the following histologic subtypes:

  * Pilocytic astrocytoma I° and variants
  * Subependymal giant cell astrocytoma I°
  * Dysembryoplastic neuroepithelial tumor I°
  * Desmoplastic infantile ganglioglioma I°
  * Ganglioglioma I° and II°
  * Pleomorphic xanthoastrocytoma II°
  * Oligodendroglioma II°
  * Oligoastrocytoma II°
  * Astrocytoma II°

    * Fibrillary astrocytoma II°
    * Protoplasmatic astrocytoma II°
    * Gemistocytic astrocytoma II°
* Children with chiasmatic-hypothalamic tumors may be eligible without histological diagnosis, if neuroradiologic findings meet unequivocal criteria for the presence of a low-grade glioma
* Primary tumor localization: intracranial and/or spinal cord

  * No diffuse intrinsic tumors of the pons, even if histologically an astrocytoma I° or II° is diagnosed

    * Exception: pontine glioma II° in neurofibromatosis type 1 (NF1) disease allowed
* Children presenting with disseminated low-grade glioma will be eligible for the study
* All eligible patients without NF1 disease receiving chemotherapy as their first nonsurgical therapy are eligible for randomization
* Children are eligible for the trial regardless of the presence of associated genetic disease: NF1 disease will be the prominent one, all children with NF1 disease are entered into the study arm III in case of an indication for nonsurgical therapy
* Patients presenting with rare intracranial neoplasms of low-grade malignancy, but nonglial origin, may be followed according to the low-grade glioma strategy, but they are not subject of this therapy trial.

  * Data from these patients may be registered to learn about those therapeutic interventions which may prove useful to these patients and to develop separate strategies in the future
  * Patients with choroid plexus papilloma should be entered into the SIOP-CPT study (Prof. Dr. J. Wolff, M.D. Anderson Cancer Center, Houston, Texas)

PATIENT CHARACTERISTICS:

* No preexisting impairments of health status, making the conduct of the study impossible or ethically unwise
* No evidence of pregnancy or lactation period
* Pregnancy has to be prevented in fertile adolescent girls during chemotherapy by reliable contraception methods (e.g., hormonal contraception)

PRIOR CONCURRENT THERAPY:

* The tumor should not be pretreated with chemotherapy or radiotherapy

  * Children treated with chemotherapy or radiotherapy prior to entering the study will be evaluated separately

    * Previous treatment with steroids is not considered a chemotherapeutic treatment
* Surgery of any type and extent allowed

  * Prior surgical resection of the tumor allowed
* Participation in another clinical study concurrently with this study (e.g., endocrinologic study) allowed provided it is not interfering with the present treatment strategy
* No other concurrent chemotherapy
* Concurrent medication for associated or other conditions (e.g., hormone replacement, anticonvulsants) that does not containing cytostatic drugs allowed

INCLUSION CRITERIA

* Age: children and adolescents up to the completion of the 18th year of life.
* Histology: low grade glioma according to ICD O Code Children with chiasmatic-hypothalamic tumors may be eligible without histological diagnosis, if neuroradiologic findings meet unequivocal criteria for the presence of a low grade glioma.
* Primary tumor localization: intracranial and/or spinal cord.
* Dissemination: Children presenting with disseminated low grade glioma will be eligible for the study.
* Associated conditions: Children are eligible for the trial regardless of the presence of associated genetic disease: Neurofibromatosis NF I will be the prominent one, all children with NF I are entered into the study arm III in case of an indication for non-surgical therapy. Other conditions like Tuberous Sclerosis etc. should be registered and their impact on the course of disease and/or therapy be followed.
* Primary tumor diagnosis: The tumor should not be pretreated with chemotherapy or radiotherapy.
* Informed consent: The patient and/or his legal guardian ( parents ) have to have declared their written informed consent to the study.

Randomization: All eligible patients without Neurofibromatosis NF I receiving chemotherapy as their fist non-surgical therapy are eligible for randomization.

EXCLUSION CRITERIA

* Primary tumor localization: diffuse intrinsic tumors of the pons, even if histologically an Astrocytoma I° or II° is diagnosed.

Exception: pontine glioma II° in NF I patients may be entered into the study.

* Special diagnosis: Patients presenting with rare intracranial neoplasms of low grade malignancy, but non-glial origin may be followed according to the low grade glioma strategy but they are not subject of this therapy trial. Their data may be registered however, to learn about those therapeutic interventions which may prove useful to these patients and to develop separate strategies in the future. Choroid plexus papilloma should be entered into the SIOP-CPT study.
* Pretreatment: Children treated with chemo- or radiotherapy prior to entering the study will be evaluated separately. (Previous treatment with steroids is not considered a chemotherapeutic treatment.)
* Preexisting impairments of health status, making the conduct of the study impossible or ethically unwise.
* Evidence of pregnancy or lactation period.

Participation in another clinical study: In case the patient participates in another clinical study simultaneously to being enrolled in the study SIOP-LGG 2004, which is not interfering with the present treatment strategy ( e.g. endocrinologic study ), this should be known to the national study chairmen.

Medication: Concomitant medication for associated or other conditions ( e.g. hormone replacement, anticonvulsants ), not containing cytostatic drugs, should be recorded, but is no exclusion criteria.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3417 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | week 24, and at 1, 3, and 5 years
Event-free survival | week 24 and at 1, 3, and 5 years
Overall survival | week 24 and at 1, 3, and 5 years

SECONDARY OUTCOMES:
Response week 24 | week 24
  radiological response to therapy (chemotherapy or radiation therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Gnekow, Study Chair — University Hospital Augsburg
Locations (13):
- Allg. Krankenhaus der Stadt Wien Universitaets-Kinderklinik, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- Aalborg Hospital, Aalborg, Denmark
- Institut Gustave Roussy, Villejuif, France
- Klinikum Augsburg, Augsburg, Germany
- Azienda Ospedaliera di Padova, Padua, Italy
- University of Tromso, Tromsø, Norway
- Children's Memorial Health Institute, Warsaw, Poland
- Hospital San Joao, Porto, Portugal
- University Children's Hospital, Zurich, Switzerland
- United Kingdom (2):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Queen's Medical Centre, Nottingham, England

REFERENCES:
- [Result] Gnekow AK, Walker DA, Kandels D, Picton S, Giorgio Perilongo, Grill J, Stokland T, Sandstrom PE, Warmuth-Metz M, Pietsch T, Giangaspero F, Schmidt R, Faldum A, Kilmartin D, De Paoli A, De Salvo GL; of the Low Grade Glioma Consortium and the participating centers. A European randomised controlled trial of the addition of etoposide to standard vincristine and carboplatin induction as part of an 18-month treatment programme for childhood (</=16 years) low grade glioma - A final report. Eur J Cancer. 2017 Aug;81:206-225. doi: 10.1016/j.ejca.2017.04.019. Epub 2017 Jun 22. PMID 28649001
- [Derived] Weiss S, Thomale UW, Schulz M, Kandels D, Schuhmann MU, El Damaty A, Krauss J, Driever PH, Witt O, Bison B, Pietsch T, Gnekow A, Simon M. Neurosurgical morbidity in pediatric supratentorial midline low-grade glioma: Results from the German LGG studies. Int J Cancer. 2023 Oct 15;153(8):1487-1500. doi: 10.1002/ijc.34615. Epub 2023 Jun 1. PMID 37260252
- [Derived] Kandels D, Pietsch T, Bison B, Warmuth-Metz M, Thomale UW, Kortmann RD, Timmermann B, Hernaiz Driever P, Witt O, Schmidt R, Gnekow AK. Loss of efficacy of subsequent nonsurgical therapy after primary treatment failure in pediatric low-grade glioma patients-Report from the German SIOP-LGG 2004 cohort. Int J Cancer. 2020 Dec 15;147(12):3471-3489. doi: 10.1002/ijc.33170. Epub 2020 Jul 11. PMID 32580249